CLINICAL TRIAL: NCT04511390
Title: Transparent Elastomeric Respirator to Protect Against Aerosol Transmission of Infectious Agents
Brief Title: Transparent Elastomeric Respirator for Aerosol-based Protection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Principal Investigator, C. Giovanni Traverso MB Bchir PhD, Assistant Professor, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020P000852
Record Dates: First submitted 2020-08-10; First posted 2020-08-13 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Personal Protective Equipment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Transparent, reusable respirator (Experimental): Transparent, reusable elastomeric respirator that has been designed to fit multiple different face sizes and shapes.
  Interventions: Device: Transparent, reusable respirator

INTERVENTIONS:
Device: Transparent, reusable respirator — A novel respirator with dual N95 filter cartridges

SUMMARY:
In times of crisis, diminishing supplies of personal protective equipment (PPE) in hospitals has forced both healthcare workers and the general population to reuse and clean PPE using anecdotal strategies which may weaken its effectiveness of preventing acquisition of airborne respiratory illnesses, such as COVID-19. There is therefore a great need to develop innovative measures to generate reusable PPE that can be safely cleaned and sterilized. A novel reusable injection molded respirator will be evaluated using qualitative and quantitative fit tests to assess overall fit and comfort.

DETAILED DESCRIPTION:
PPE is the last line of defense in the hierarchy of controls to prevent the spread of airborne transmissible infections. There are many varieties of respirators including quarter-mask, half mask, and full facepiece respirators that filter 95, 99, or 100% of airborne particles. The elastomeric half mask respirators (EHMRs), in particular, have several advantages over commonly used N95 FFRs. Firstly, EHMRs may be cleaned, disinfected, and reused unlike FFRs that are normally discarded after a single use. EHMRs may be transparent as a result of material choice and will allow for visualization of the mouth. Lastly, they have been shown to properly fit faces after multiple rounds of decontamination.

Some disadvantages of EHMRs include the requirement to disinfect and reinspect the quality of components on the respirator by a qualified individual for proper function, as well as manual exchange of filter components. Notwithstanding, it has been found that fit testing and training to use EHMRs for healthcare personnel is not significantly different than N95 respirators and that EHMR may serve as a suitable alternative to disposable N95 respirators during public health emergencies. Furthermore, a 2018 consensus report from the National Academies of Engineering, Science, and Medicine recommended that the durability and reusability of elastomeric respirators made them desirable for stockpiling for emergencies.

A new transparent elastomeric respirator has been developed that can maintain respirator integrity after decontamination and fits many people with different face sizes and shapes. Fit testing of the respirator will be performed using an OSHA-approved testing method.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers that have undergone successful fit test with N95 FFR within 1 year of the trial

Exclusion Criteria:

* Facial hair

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-25 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Success of fit testing | 30 minutes
  Successful fit testing using an Occupational Safety and Health Administration (OSHA)-approved testing method testing method

SECONDARY OUTCOMES:
User experience | 30 minutes
  User experience with fit, breathability and filter replacement will be assessed based on a Likert scale through a post-fit test questionnaire

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided